CLINICAL TRIAL: NCT01061073
Title: Evaluation of the Efficacy of Tamsulosin (Alpha Blockers) Compared to Phloroglucinol in Improving JJ Ureteral Stent Tolerance. A Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Pr IRANI - principal investigator, CHU DE POITIERS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JJ Alpha 2009
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Non-oncological Indication to Ureteral Stenting
MeSH Terms: interventions — 1,3,5-benzenetriol, 1,3,5-trimethoxybenzene drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omexel (Experimental)
  Interventions: Drug: Omexel
- spasfon (Active Comparator)
  Interventions: Drug: spasfon

INTERVENTIONS:
Drug: Omexel
  Arms: Omexel
Drug: spasfon
  Arms: spasfon

SUMMARY:
JJ ureteral stent represents an advance in the management of the upper urinary tract obstruction as it allows the patient to resume his activities although he is stented between the kidney and the bladder.

However, in many cases, this JJ stent is not well tolerated and can even be unbearable.

This trial evaluates the benefit of tamsulosin (an alpha-blocker) in improving the tolerance of JJ stents compared to low-doses of phloroglucinol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 or more.
2. Non-oncological indication to ureteral stenting
3. Informed written consent

Exclusion Criteria:

1 Any contra-indication to Tamsulosin or phloroglucinol (renal or hepatic insufficiency, allergy) 2. Pregnancy 3. Patients already treated with alpha blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the benefit of alpha-blockers (Tamsulosin, group A) compared to phloroglucinol (Spasfon®, group B) as regards patients tolerance to JJ stents | 1 month treatment

SECONDARY OUTCOMES:
incidence of complications | after 1 month treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital - 2 rue de la Milétrie, Poitiers, France